CLINICAL TRIAL: NCT03141437
Title: Patient-Centered Decision Counseling for Women at Risk of Cancer-Related Infertility: Efficacy Study and Comparative-Effectiveness Randomized Trial
Brief Title: Decision Aid Website in Helping to Make Decisions About Fertility in Participants With Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-0758; NCI-2018-01208 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0758 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); UG1CA189823 (NIH)
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasm; Colorectal Neoplasm; Female Reproductive System Neoplasm; Health Care Provider; Lymphoma; Plasma Cell Myeloma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Genital Neoplasms, Female; Lymphoma; Multiple Myeloma | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (standard of care) (Active Comparator): Participants receive standard of care including education materials about fertility preservation from the Livestrong organization and a referral for fertility preservation, if requested.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Questionnaire Administration
- Arm II (standard of care, decision-making website) (Experimental): Participants receive standard of care as in Arm I. Participants also use the decision-making the website.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Internet-Based Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Other: Educational Intervention — Receive educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Internet-Based Intervention — Use decision-making website
  Arms: Arm II (standard of care, decision-making website)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a decision aid website works in helping to make decisions about fertility in participants with cancer. Decision aid websites that provide information about fertility preservation (maintaining your ability to have children of your own after cancer treatment) may help participants with cancer make fertility-preservation decisions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the effect of the Pathways to Fertility patient decision aid website (DA website) with women of reproductive age seen at the MD Anderson Oncofertility Service, in terms of improving patients' decisional conflict. (Part 1) II. To assess the effect of a multicomponent oncofertility decision support intervention (multicomponent DS intervention) compared to usual care with women of reproductive age at selected MD Anderson Houston Area Locations (HALs) on patients' decisional conflict. (Part 2)

SECONDARY OBJECTIVES:

I. To assess patients' decision-making process (e.g., preparation for decision making, decision self-efficacy, satisfaction) and decision quality (e.g., fertility preservation knowledge, clarity of patients' values, and congruence of preferences with the decision and/or treatment received). (Part 1) II. To assess patients' decision-making process (e.g., preparation for decision making, decision self-efficacy, satisfaction) and decision quality (e.g., fertility preservation knowledge, clarity of patients' values, and congruence of preferences with the decision about whether to accept fertility preservation referral and/or fertility preservation treatment). (Part 2)

EXPLORATORY OBJECTIVES:

I. To explore the acceptability of the DA website (e.g., length, clarity, ease of use) and feasibility of the research methods (e.g., preferences for viewing at home versus at the clinic, timing of viewing, website usage, recommendations for improvement), in preparation for future planned dissemination and implementation studies. (Part 1) II. To explore the feasibility of the multicomponent DS intervention and research methods (e.g., clinician's perspectives of the educational session and referral process, website usage, rates of referrals, recommendations for improving the intervention and referral process) as delivered in the HALs oncology clinics, in preparation for future planned dissemination and implementation studies. (Part 2)

OUTLINE:

PART 1: Participants review decision aid website and complete questionnaires to help researchers learn the website's effect.

PART 2: Participants are randomized into 1 of 2 arms.

ARM I: Participants receive standard of care including education materials about fertility preservation from the Livestrong organization and a referral for fertility preservation, if requested.

ARM II: Participants receive standard of care as in Arm I. Participants also use the decision-making the website.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast tumor, female genital system tumor, colorectal tumor, and/or lymphoma/myeloma
* At risk for cancer-related infertility, as assessed by their clinician(s), including the oncofertility specialist
* Must be able to speak, read, and write English
* Must have internet access and a valid email address
* Have not previously viewed the Pathways decision aid
* For clinical provider participants: Clinical provider at a Houston Area Location of MD Anderson assigned to the intervention

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-04-23 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Patients' decisional conflict (Part 1) | Up to 2 months
  Will assess the effect of the Pathways to Fertility patient decision aid website (DA website) with women of reproductive age seen at the MD Anderson Oncofertility Service, in terms of improving patients' decisional conflict.
Patients' decisional conflict (Part 2) | Up to 2 months
  Will assess the effect of a multicomponent oncofertility decision support intervention (multicomponent DS intervention) compared to usual care with women of reproductive age at selected MD Anderson Houston Area Locations (HALs) on patients' decisional conflict.

SECONDARY OUTCOMES:
Patients' decision-making process (Part 1) | Up to 2 months
  Will assess patients' decision-making process (e.g., preparation for decision making, decision self-efficacy, satisfaction) and decision quality (e.g., fertility preservation knowledge, clarity of patients' values, and congruence of preferences with the decision and/or treatment received).
Patients' decision-making process (Part 2) | Up to 2 months
  Will assess patients' decision-making process (e.g., preparation for decision making, decision self-efficacy, satisfaction) and decision quality (e.g., fertility preservation knowledge, clarity of patients' values, and congruence of preferences with the decision about whether to accept fertility preservation referral and/or fertility preservation treatment).

OTHER OUTCOMES:
Acceptability of the decision aid website (Part 1) | Up to 2 months
  Will explore the acceptability of the DA website (e.g., length, clarity, ease of use) and feasibility of the research methods (e.g., preferences for viewing at home versus at the clinic, timing of viewing, website usage, recommendations for improvement), in preparation for future planned dissemination and implementation studies.
Feasibility of the multicomponent DS intervention and research methods (Part 2) | Up to 2 months
  Will explore the feasibility of the multicomponent DS intervention and research methods (e.g., clinician's perspectives of the educational session and referral process, website usage, rates of referrals, recommendations for improving the intervention and referral process) as delivered in the HALs oncology clinics, in preparation for future planned dissemination and implementation studies.

CONTACTS AND LOCATIONS:
Overall Officials: Terri L Woodard, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Woodard TL, Hoffman AS, Crocker LC, Holman DA, Hoffman DB, Ma J, Bassett RL Jr, Leal VB, Volk RJ. Pathways: patient-centred decision counselling for women at risk of cancer-related infertility: a protocol for a comparative effectiveness cluster randomised trial. BMJ Open. 2018 Feb 21;8(2):e019994. doi: 10.1136/bmjopen-2017-019994. PMID 29467138
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org